CLINICAL TRIAL: NCT05378204
Title: Prospective and Multicentric Study Evaluating DNA Double-strand Breaks (DSBs) REpair Factors (POLQ, Shieldin Complex and 53BP1) Expression as Biomarker of PARP Inhibitor Resistance in Patients With Deleterious Germline Mutation in BRCA 1/2 and HER2-negative, Metastatic or Locally Advanced Breast Cancer.
Brief Title: Study Evaluating DNA Double-strand Breaks (DSBs) REpair Factors (POLQ, Shieldin Complex and 53BP1) Expression as Biomarker of PARP Inhibitor Resistance in Patients With Deleterious Germline Mutation in BRCA 1/2 and HER2-negative, Metastatic or Locally Advanced Breast Cancer.
Acronym: REPARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21 SEIN 09
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Germline BRCA mutation; PARP inhibitor; Biomarkers; POLQ; Polθ; Shieldin complex; 53BP1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with breast cancer (Other): Patients With Deleterious Germline Mutation in BRCA 1/2 and HER2-negative, Metastatic or Locally Advanced Breast Cancer.
  Interventions: Other: Main study:; Other: Sub-study:

INTERVENTIONS:
Other: Main study: — For each included patient, tumor biopsy specimen and blood samples will be collected at baseline visit (before the first dose of PARPi treatment).
  During the treatment period: blood samples will be scheduled every 8 weeks (i.e. 2 cycles).
  At the time of progression: tumor biopsy and blood samples will be collected.
Other: Sub-study: — For each included patient, tumor biopsy specimen and blood samples will be collected as soon as possible after progression (before initiation of the post PARPi anti-tumoral treatment).

SUMMARY:
The purpose of this study is to assess whether expression of not only POLQ/Polθ, but also Shieldin complex and/or 53BP1 are correlated with primary and/or acquired resistance to PARPi (Poly(ADP-Ribose) Polymerases inhibitors) in a sub-population of locally advanced or metastatic breast cancer patients and vary regarding type and location of gBRCA1/2 mutations.

This translational research program is composed of two multicentric, non-randomized prospective studies in patients with HER2-negative locally advanced or metastatic breast cancer:

* The main study concerns 80 patients eligible for PARPi (according to the investigators).PARPi treatments (talazoparib or olaparib) will be administered and dosed according to the standard of care administration.
* The sub-study concerns 40 patients in progression disease under PARPi alone.

For each included patient in the main study or sub-study, tumor biopsy specimen and blood samples will be collected at different times during the study.

ELIGIBILITY:
MAIN STUDY

INCLUSION CRITERIA:

1. Women (or men) aged ≥ 18 years with histologically proven breast cancer
2. Metastatic relapse or locally advanced breast cancer
3. No-HER2 overexpression or amplification
4. Triple-negative (defines as ER<1%, PR<1% and HER2-negative as per ASCO CAP guidelines) or hormone receptor positive (defines as ER and/or PR ≥ 1%) breast cancer
5. Patients with metastases that can be biopsied except bone metastases. At baseline, if patients already have an archived biopsy from a secondary or a primary site (if stage IV) of their current disease, this material can be used for the study, provided that, it was collected within 3 months prior enrollment and a frozen and a FFPE sample are both available for research
6. ECOG Performance Status ≤ 2
7. Patients must have measurable or evaluable disease according to RECIST v1.1
8. Patient with deleterious germline BRCA 1 and/or 2 mutation, eligible for PARP inhibitor therapy (olaparib or talazoparib), according each investigator
9. Any number of prior lines therapy are allowed
10. Current treatment with PARP inhibitor not yet started
11. Women should be post-menopaused or willing to accept the use of an effective contraceptive regimen during the treatment period by PARP inhibitor
12. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
13. Patient affiliated to a Social Health Insurance in France

NON-INCLUSION CRITERIA:

1. Abnormal coagulation contraindicating biopsy
2. Bone metastases when this is the only site of biopsiable disease
3. Patients with all target in a previously irradiated region, except if clear progression has been observed prior to study in at least one of them
4. Patients with known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
5. Patients with known untreated CNS metastases and/or carcinomatous meningitis
6. Patients with a known history of Human Immunodeficiency Virus (HIV)
7. Patients with known active Hepatitis B or C
8. Patients should not be on any other anti-cancer therapy (chemotherapy, endocrine therapy, immunotherapy, tailored therapy or alternative investigational therapy)
9. Patient pregnant, or breast-feeding
10. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
11. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

SUB-STUDY

INCLUSION CRITERIA:

1. Women (or men) aged ≥ 18 years with histologically proven breast cancer
2. Metastatic relapse or locally advanced breast cancer
3. No-HER2 overexpression or amplification
4. Triple-negative (defines as ER<1%, PR<1% and HER2-negative as per ASCO CAP guidelines) or hormone receptor positive (defines as ER and or PR ≥ 1%) breast cancer
5. Patients with metastases that can be biopsied except bone metastases
6. ECOG Performance Status ≤ 2
7. Patients, with deleterious germline BRCA 1 and/or 2, in progression under PARPi alone (talazoparib or olaparib)
8. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
9. Patient affiliated to a Social Health Insurance in France

NON-INCLUSION CRITERIA:

1. Abnormal coagulation contraindicating biopsy
2. Bone metastases when this is the only site of biopsiable disease
3. Patient pregnant, or breast-feeding
4. Patients with a known history of Human Immunodeficiency Virus (HIV)
5. Patients with known active Hepatitis B or C
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
7. Patients already participating in the main REPARP study
8. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Main study: the primary endpoint is the Area under the Receiver Operating Characteristic Curve (ROC Curve) of POLQ expression to identify patients presenting progressive disease or death at 6 months under PARPi alone (primary resistance). | 6 months for each patient
  Progression will be determined using RECIST v1.1 criteria.
Sub-study: the primary end point is the rate of patients presenting loss of Shieldin complex and/or 53BP1. | 1 month for each patient

SECONDARY OUTCOMES:
Main study: Progression-Free Survival defined as the time from inclusion until progression according to RECIST v1.1 criteria or death from any cause, whichever occurs first. | 12 months for each patient
Main study: Objective Response (i.e. complete or partial response) defined using RECIST v1.1 criteria. | 12 months for each patient
Main study: Duration Of Response defined as the time from initial objective response until progression according to RECIST v1.1 criteria or death from any cause. | 12 months for each patient
Sub-study: expression of the Shieldin complex and 53BP1. | 1 month for each patient

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - CHU de LIMOGES, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre de Cancerologie Du Grand Montpellier, Montpellier
  - Institut Regional Du Cancer de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - Hopital Pitie Salpetriere, Paris
  - Hopital Saint Louis, Paris
  - Hopital Tenon, Paris
  - INSTITUT CURIE - Site de Paris, Paris
  - CENTRE ARMORICAIN DE RADIOTHERAPIE, IMAGERIE MEDICALE ET ONCOLOGIE - Hôpital privé des Côtes d'Armor, Plérin
  - Chu de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Chu Saint Etienne, Saint-Etienne
  - INSTITUT DE CANCEROLOGIE DE L'OUEST St-Herblain, Saint-Herblain
  - IUCT-O, Toulouse
  - Chru de Tours, Tours
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif